CLINICAL TRIAL: NCT01055054
Title: Analysis Bariatric Surgery Data
Brief Title: Bariatric Surgery Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM1587
Record Dates: First submitted 2010-01-20; First posted 2010-01-25 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Morbid
Keywords: bariatrics
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Periodic analyses of our extensive database with regards to different surgical procedures for severe obesity and different obesity co-morbidities will be of benefit to our severely obese patients as well as to others world-wide.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of morbid obesity
* Have undergone a bariatric surgical procedure at the VCU Medical Center

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone bariatric surgical procedures at the Virginia Commonwealth University (VCU) Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 1980-07-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
weight loss | 1 year, 5 years

SECONDARY OUTCOMES:
surgical mortality | 90 day post-surgery
surgical morbidity | 90 day post-surgery
resolution of co-morbidities | 1 year, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Campos, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU Health Systems, Richmond, Virginia, United States

REFERENCES:
- [Result] Sugerman HJ, Fairman RP, Baron PL, Kwentus JA. Gastric surgery for respiratory insufficiency of obesity. Chest. 1986 Jul;90(1):81-6. doi: 10.1378/chest.90.1.81. PMID 3720390
- [Result] Sugerman HJ, Starkey JV, Birkenhauer R. A randomized prospective trial of gastric bypass versus vertical banded gastroplasty for morbid obesity and their effects on sweets versus non-sweets eaters. Ann Surg. 1987 Jun;205(6):613-24. doi: 10.1097/00000658-198706000-00002. PMID 3296971
- [Result] Sugerman HJ, Baron PL, Fairman RP, Evans CR, Vetrovec GW. Hemodynamic dysfunction in obesity hypoventilation syndrome and the effects of treatment with surgically induced weight loss. Ann Surg. 1988 May;207(5):604-13. doi: 10.1097/00000658-198805000-00015. PMID 3377570
- [Result] Sugerman HJ, Londrey GL, Kellum JM, Wolf L, Liszka T, Engle KM, Birkenhauer R, Starkey JV. Weight loss with vertical banded gastroplasty and Roux-Y gastric bypass for morbid obesity with selective versus random assignment. Am J Surg. 1989 Jan;157(1):93-102. doi: 10.1016/0002-9610(89)90427-3. PMID 2910132
- [Result] Sugerman HJ, Fairman RP, Sood RK, Engle K, Wolfe L, Kellum JM. Long-term effects of gastric surgery for treating respiratory insufficiency of obesity. Am J Clin Nutr. 1992 Feb;55(2 Suppl):597S-601S. doi: 10.1093/ajcn/55.2.597s. PMID 1733136
- [Result] Sanyal AJ, Sugerman HJ, Kellum JM, Engle KM, Wolfe L. Stomal complications of gastric bypass: incidence and outcome of therapy. Am J Gastroenterol. 1992 Sep;87(9):1165-9. PMID 1519574
- [Result] Sugerman HJ, Sugerman EL, Wolfe L, Kellum JM Jr, Schweitzer MA, DeMaria EJ. Risks and benefits of gastric bypass in morbidly obese patients with severe venous stasis disease. Ann Surg. 2001 Jul;234(1):41-6. doi: 10.1097/00000658-200107000-00007. PMID 11460821
- [Result] DeMaria EJ, Sugerman HJ, Kellum JM, Meador JG, Wolfe LG. Results of 281 consecutive total laparoscopic Roux-en-Y gastric bypasses to treat morbid obesity. Ann Surg. 2002 May;235(5):640-5; discussion 645-7. doi: 10.1097/00000658-200205000-00005. PMID 11981209
- [Result] DeMaria EJ, Schweitzer MA, Kellum JM, Meador J, Wolfe L, Sugerman HJ. Hand-assisted laparoscopic gastric bypass does not improve outcome and increases costs when compared to open gastric bypass for the surgical treatment of obesity. Surg Endosc. 2002 Oct;16(10):1452-5. doi: 10.1007/s00464-001-8321-5. Epub 2002 Jun 14. PMID 12063573
- [Result] Kothari SN, DeMaria EJ, Sugerman HJ, Kellum JM, Meador J, Wolfe L. Lap-band failures: conversion to gastric bypass and their preliminary outcomes. Surgery. 2002 Jun;131(6):625-9. doi: 10.1067/msy.2002.124879. PMID 12075174
- [Result] Sugerman HJ, Sugerman EL, DeMaria EJ, Kellum JM, Kennedy C, Mowery Y, Wolfe LG. Bariatric surgery for severely obese adolescents. J Gastrointest Surg. 2003 Jan;7(1):102-108. doi: 10.1016/S1091-255X(02)00125-7. PMID 12559191
- [Result] Sugerman HJ, Wolfe LG, Sica DA, Clore JN. Diabetes and hypertension in severe obesity and effects of gastric bypass-induced weight loss. Ann Surg. 2003 Jun;237(6):751-6; discussion 757-8. doi: 10.1097/01.SLA.0000071560.76194.11. PMID 12796570
- [Result] Fernandez AZ Jr, DeMaria EJ, Tichansky DS, Kellum JM, Wolfe LG, Meador J, Sugerman HJ. Experience with over 3,000 open and laparoscopic bariatric procedures: multivariate analysis of factors related to leak and resultant mortality. Surg Endosc. 2004 Feb;18(2):193-7. doi: 10.1007/s00464-003-8926-y. Epub 2003 Dec 29. PMID 14691697
- [Result] Fernandez AZ Jr, Demaria EJ, Tichansky DS, Kellum JM, Wolfe LG, Meador J, Sugerman HJ. Multivariate analysis of risk factors for death following gastric bypass for treatment of morbid obesity. Ann Surg. 2004 May;239(5):698-702; discussion 702-3. doi: 10.1097/01.sla.0000124295.41578.ab. PMID 15082974
- [Result] Sugerman HJ, DeMaria EJ, Kellum JM, Sugerman EL, Meador JG, Wolfe LG. Effects of bariatric surgery in older patients. Ann Surg. 2004 Aug;240(2):243-7. doi: 10.1097/01.sla.0000133361.68436.da. PMID 15273547
- [Result] Bond DS, Evans RK, Wolfe LG, Meador JG, Sugerman HJ, Kellum JM, Demaria EJ. Impact of self-reported physical activity participation on proportion of excess weight loss and BMI among gastric bypass surgery patients. Am Surg. 2004 Sep;70(9):811-4. PMID 15481300
- [Result] Tichansky DS, DeMaria EJ, Fernandez AZ, Kellum JM, Wolfe LG, Meador JG, Sugerman HJ. Postoperative complications are not increased in super-super obese patients who undergo laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2005 Jul;19(7):939-41. doi: 10.1007/s00464-004-8929-3. Epub 2005 May 5. PMID 15920681
- [Result] Carmody BJ, Sugerman HJ, Kellum JM, Jamal MK, Johnson JM, Carbonell AM, Maher JW, Wolfe LG, DeMaria EJ. Pulmonary embolism complicating bariatric surgery: detailed analysis of a single institution's 24-year experience. J Am Coll Surg. 2006 Dec;203(6):831-7. doi: 10.1016/j.jamcollsurg.2006.08.020. Epub 2006 Oct 25. PMID 17116551
- [Result] Carbonell AM, Wolfe LG, Meador JG, Sugerman HJ, Kellum JM, Maher JW. Does diabetes affect weight loss after gastric bypass? Surg Obes Relat Dis. 2008 May-Jun;4(3):441-4. doi: 10.1016/j.soard.2007.10.001. Epub 2007 Dec 11. PMID 18065289
- [Result] Ali MR, Tichansky DS, Kothari SN, McBride CL, Fernandez AZ Jr, Sugerman HJ, Kellum JM, Wolfe LG, DeMaria EJ. Validation that a 1-year fellowship in minimally invasive and bariatric surgery can eliminate the learning curve for laparoscopic gastric bypass. Surg Endosc. 2010 Jan;24(1):138-44. doi: 10.1007/s00464-009-0550-z. Epub 2009 Jun 11. PMID 19517173
- [Result] Evans RK, Bond DS, Demaria EJ, Wolfe LG, Meador JG, Kellum JM. Initiation and progression of physical activity after laparoscopic and open gastric bypass surgery. Surg Innov. 2004 Dec;11(4):235-9. doi: 10.1177/155335060401100406. PMID 15756392
- [Result] Johnson JM, Maher JW, DeMaria EJ, Downs RW, Wolfe LG, Kellum JM. The long-term effects of gastric bypass on vitamin D metabolism. Ann Surg. 2006 May;243(5):701-4; discussion 704-5. doi: 10.1097/01.sla.0000216773.47825.c1. PMID 16633006
- [Result] Bond DS, Evans RK, DeMaria E, Wolfe L, Meador J, Kellum J, Maher J, Warren BJ. Physical activity and quality of life improvements before obesity surgery. Am J Health Behav. 2006 Jul-Aug;30(4):422-34. doi: 10.5555/ajhb.2006.30.4.422. PMID 16787132
- [Result] Jamal MK, DeMaria EJ, Johnson JM, Carmody BJ, Wolfe LG, Kellum JM, Meador JG. Impact of major co-morbidities on mortality and complications after gastric bypass. Surg Obes Relat Dis. 2005 Nov-Dec;1(6):511-6. doi: 10.1016/j.soard.2005.08.010. Epub 2005 Oct 27. PMID 16925280
- [Result] Jamal MK, DeMaria EJ, Johnson JM, Carmody BJ, Wolfe LG, Kellum JM, Meador JG. Insurance-mandated preoperative dietary counseling does not improve outcome and increases dropout rates in patients considering gastric bypass surgery for morbid obesity. Surg Obes Relat Dis. 2006 Mar-Apr;2(2):122-7. doi: 10.1016/j.soard.2006.01.009. PMID 16925335
- [Result] Bond DS, Evans RK, DeMaria EJ, Wolfe LG, Meador JG, Kellum JM, Maher JW. Physical activity stage of readiness predicts moderate-vigorous physical activity participation among morbidly obese gastric bypass surgery candidates. Surg Obes Relat Dis. 2006 Mar-Apr;2(2):128-32. doi: 10.1016/j.soard.2006.01.007. Epub 2006 Mar 3. PMID 16925336
- [Result] DeMaria EJ, Portenier D, Wolfe L. Obesity surgery mortality risk score: proposal for a clinically useful score to predict mortality risk in patients undergoing gastric bypass. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):134-40. doi: 10.1016/j.soard.2007.01.005. PMID 17386394
- [Result] Lee S, Carmody B, Wolfe L, Demaria E, Kellum JM, Sugerman H, Maher JW. Effect of location and speed of diagnosis on anastomotic leak outcomes in 3828 gastric bypass cases. J Gastrointest Surg. 2007 Jun;11(6):708-13. doi: 10.1007/s11605-007-0085-3. PMID 17562118
- [Result] Lee SD, Khouzam MN, Kellum JM, DeMaria EJ, Meador JG, Wolfe LG, Maher JW. Selective, versus routine, upper gastrointestinal series leads to equal morbidity and reduced hospital stay in laparoscopic gastric bypass patients. Surg Obes Relat Dis. 2007 Jul-Aug;3(4):413-6. doi: 10.1016/j.soard.2007.04.006. Epub 2007 Jun 12. PMID 17567540
- [Result] Evans RK, Bond DS, Wolfe LG, Meador JG, Herrick JE, Kellum JM, Maher JW. Participation in 150 min/wk of moderate or higher intensity physical activity yields greater weight loss after gastric bypass surgery. Surg Obes Relat Dis. 2007 Sep-Oct;3(5):526-30. doi: 10.1016/j.soard.2007.06.002. PMID 17903772
- [Result] Maher JW, Martin Hawver L, Pucci A, Wolfe LG, Meador JG, Kellum JM. Four hundred fifty consecutive laparoscopic Roux-en-Y gastric bypasses with no mortality and declining leak rates and lengths of stay in a bariatric training program. J Am Coll Surg. 2008 May;206(5):940-4; discussion 944-5. doi: 10.1016/j.jamcollsurg.2007.12.043. Epub 2008 Mar 24. PMID 18471729
- [Result] Yuan X, Martin Hawver LR, Ojo P, Wolfe LM, Meador JG, Kellum JM, Maher JW. Bariatric surgery in Medicare patients: greater risks but substantial benefits. Surg Obes Relat Dis. 2009 May-Jun;5(3):299-304. doi: 10.1016/j.soard.2008.08.018. Epub 2008 Aug 30. PMID 18996764
- [Result] Bond DS, Phelan S, Wolfe LG, Evans RK, Meador JG, Kellum JM, Maher JW, Wing RR. Becoming physically active after bariatric surgery is associated with improved weight loss and health-related quality of life. Obesity (Silver Spring). 2009 Jan;17(1):78-83. doi: 10.1038/oby.2008.501. Epub 2008 Nov 6. PMID 18997679
- [Result] Maher JW, Bakhos W, Nahmias N, Wolfe LG, Meador JG, Baugh N, Kellum JM. Drain amylase levels are an adjunct in detection of gastrojejunostomy leaks after Roux-en-Y gastric bypass. J Am Coll Surg. 2009 May;208(5):881-4; discussion 885-6. doi: 10.1016/j.jamcollsurg.2008.12.022. Epub 2009 Mar 26. PMID 19476853
- [Result] Chikunguwo SM, Wolfe LG, Dodson P, Meador JG, Baugh N, Clore JN, Kellum JM, Maher JW. Analysis of factors associated with durable remission of diabetes after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2010 May-Jun;6(3):254-9. doi: 10.1016/j.soard.2009.11.003. Epub 2009 Nov 10. PMID 20303324
- [Result] Kellum JM, Chikunguwo SM, Maher JW, Wolfe LG, Sugerman HJ. Long-term results of malabsorptive distal Roux-en-Y gastric bypass in superobese patients. Surg Obes Relat Dis. 2011 Mar-Apr;7(2):189-93. doi: 10.1016/j.soard.2010.08.018. Epub 2010 Oct 11. PMID 21145293
- [Result] Browning MG, Baugh NG, Wolfe LG, Kellum JK, Maher JW, Evans RK. Evaluation of pre- and postoperative physical activity participation in laparoscopic gastric banding patients. Obes Surg. 2014 Nov;24(11):1981-6. doi: 10.1007/s11695-014-1283-1. PMID 24831460
- [Result] Browning MG, Khoraki J, DeAntonio JH, Mazzini G, Mangino MJ, Siddiqui MS, Wolfe LG, Campos GM. Protective effect of black relative to white race against non-alcoholic fatty liver disease in patients with severe obesity, independent of type 2 diabetes. Int J Obes (Lond). 2018 Apr;42(4):926-929. doi: 10.1038/ijo.2017.309. Epub 2017 Dec 21. PMID 29437160
- [Result] Khoraki J, Mazzini GS, Shah AS, Del Prado PAR, Wolfe LG, Campos GM. Early small bowel obstruction after laparoscopic gastric bypass: a surgical emergency. Surg Obes Relat Dis. 2018 Aug;14(8):1118-1125. doi: 10.1016/j.soard.2018.05.009. Epub 2018 May 23. PMID 29945755
- [Result] Pessoa BM, Browning MG, Mazzini GS, Wolfe L, Kaplan A, Khoraki J, Campos GM. Factors Mediating Type 2 Diabetes Remission and Relapse after Gastric Bypass Surgery. J Am Coll Surg. 2020 Jan;230(1):7-16. doi: 10.1016/j.jamcollsurg.2019.09.012. Epub 2019 Oct 28. PMID 31672669
- [Result] Mazzini GS, Khoraki J, Browning MG, Pessoa BM, Wolfe LG, Campos GM. Population Diversity Challenge the External Validity of the European Randomized Controlled Trials Comparing Laparoscopic Gastric Bypass and Sleeve Gastrectomy. Obes Surg. 2020 Mar;30(3):992-1000. doi: 10.1007/s11695-019-04247-y. PMID 31768868